CLINICAL TRIAL: NCT06111417
Title: Use of an Ultra-rapid BRCA1/2 Status Screening Test in Diagnostic and Theranostic Indication: Performance and Interest for Patients and Practitioners
Acronym: TURBO
Status: Recruiting | Type: Observational
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A02176-39
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: BRCA 1/2; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard arm: Analysis carried out using the gold standard with BRCA1/2 results provided on average in 2 months for the theranostic analysis and 3 months for the "standard" analysis + ultrafast BRCA1/2 test (nanopore test) with no communication of results to the patient at 1-2 weeks.
  Interventions: Other: Questionnaires
- Experimental arm: Analysis carried out using the gold standard with BRCA1/2 results provided in an average of 2 months for the theranostic analysis and 3 months for the "standard" analysis + ultra-rapid BRCA1/2 test (nanopore test) with results communicated to the patient in 1-2 weeks. This communication will be accompanied by the necessary explanations to enable the patient to understand that this is a preliminary result and that only the gold standard will constitute a definitive result.
  Interventions: Other: Questionnaires; Other: Communication of the results of the BRCA1/2 ultra rapid test

INTERVENTIONS:
Other: Questionnaires — 3 questionnaires to allowed to assess satisfaction and acceptance of the nanopore ultrafast test by practitioners and anxiety of results by patients :
  * STAI-Y (State-Trait Anxiety Inventory)
  * Patient's Questionnaire
  * Practitioner's questionnaire
Other: Communication of the results of the BRCA1/2 ultra rapid test — Communication of the results of the BRCA1/2 ultra rapid test during a consultation 1 to 2 weeks after the test
  Groups: Experimental arm

SUMMARY:
The time taken to obtain the results of germline mutations in BRCA1 and BRCA2 has become a major issue in adapting the therapeutic management of patients, particularly those with breast cancer.

The time taken to obtain the results of BRCA1/2 tests in routine laboratories with a view to personalised treatment can range from a few weeks to a few months. The waiting time required to obtain results is likely to cause stress and anxiety in cancer patients. The investigators hypothesise that ultra-rapid testing can reduce anxiety about patients' genetic status and improve their mental well-being.

The main objective of this project is to compare the results obtained with an ultra-fast kit developed by O.N.T with those obtained with the current gold standard, NGS sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Indication for oncogenetic consultation with a wide panel test including BRCA1/2 (gold standard) as part of the standard theranostic and diagnostic management of breast cancer.
* The patient agrees to take part in the study, to follow all the study procedures and to complete the questionnaires sent during the consultation or by email.
* Diagnosis of the disease ≤ 6 months
* The patient must be affiliated to the social security system.

Exclusion Criteria:

* Concomitant disorder or condition likely to compromise understanding of study information or completion of questionnaires
* Patients who do not have an email address and/or do not have internet access or tools to connect to the internet
* Women who are pregnant, may become pregnant or are breast-feeding
* Persons deprived of their liberty or under guardianship (including curatorship)
* Inability to undergo trial monitoring for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer with an indication for theranostic BRCA1/2 analysis or diagnostic BRCA1/2 analysis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-09-12 (Estimated); Study Completion 2026-09-12 (Estimated)

PRIMARY OUTCOMES:
Compare the results obtained with an ultra-rapid kit BRCA1/2 with those obtained with the current gold standard, by checking the sensitivity, specificity and the rate of patients correctly classified for BRCA1 and 2 status | During 2 months
  The main objective will be to determine the rate of misclassified patients by pooling the 2 arms, false positives and false negatives.
  * True positives (VP) : patients presenting a BRCA 1 or 2 mutation with the ultrafast BRCA1/2 test and the gold standard.
  * False positives (FP) : patients with a BRCA 1 or 2 mutation using the BRCA1/2 ultrafast test and no BRCA 1 or 2 mutation using the gold standard.
  * True negatives (VN) : patients with no BRCA 1 or 2 mutation using the BRCA1/2 ultrafast test and the gold standard.
  * False negatives (FN) : patients without a BRCA 1 or 2 mutation using the BRCA1/2 ultrafast test and with a BRCA 1 or 2 mutation using the standard test.
  WELL classified = VP + VN, poorly classified= FP+ FN FPs will generate anxiety, and FNs will lead to a loss of chance for patients if the ultrafast BRCA1/2 test (nanopore test) is used exclusively instead of the gold standard. The overall number of misclassified patients must therefore be limited.

SECONDARY OUTCOMES:
Evaluate the sensitivity and specificity of the ultra-rapid BRCA1/2 test | During 2 months
  Evaluate the sensitivity and specificity of the ultra-rapid BRCA1/2 test (nanopore test) compared with the standard BRCA1/2 test (gold standard).
To assess the impact on patients' mental well-being (anxiety or reassurance) using the State-Trait Anxiety Questionnaire (STAI-Y) | During 2 months
  Anxiety will be assessed in each arm using the State-Trait Anxiety Questionnaire (STAI-Y) at 4 different time points:
  * After the patient has not objected to taking part in the TURBO study at the first consultation (before randomization);
  * 1-2 weeks after inclusion. The questionnaire will be e-mailed to patients. The questionnaire must be completed before the results of the BRCA1/2 ultrafast test (nanopore test) are communicated to patients in the experimental group.
  * 4 weeks after inclusion. The questionnaire will be sent by email.
  * 8 - 12 weeks after inclusion, during the consultation for the communication of test results with the gold standard, before the communication of results.
Evaluate clinician satisfaction with satisfaction scale used in genetic counselling | During 2 months
  Clinician satisfaction (oncogeneticist and oncologist) and acceptance of the BRCA1/2 ultrafast test (nanopore test) will be evaluated in both arms using a questionnaire to assess clinician satisfaction at 2 different times for each practitioner involved in patient follow-up:
  * When the first patient is unopposed;
  * At the last patient's discharge.
Evaluate patient satisfaction used in genetic counselling | During 2 months
  Patient satisfaction will be assessed in both arms using a satisfaction scale used in genetic counselling at two different times:
  * After the patient has made no objection to participating in the TURBO study during the first consultation (before randomization);
  * 8 - 12 weeks after inclusion, before the consultation for the gold standard test results.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Georges-François Leclerc, Dijon
  - Institut Rafaël, Levallois-Perret

IPD SHARING:
Plan to Share IPD: No